CLINICAL TRIAL: NCT00872586
Title: A Randomized, Double-blind, Double-dummy, Multicenter Clinical Trial to Evaluate the Additional Efficacy and Safety of Olmesartan Medoxomil 20mg / Hydrochlorothiazide 12.5mg in the Treatment of Chinese Patients With Mild to Moderate Essential Hypertension, Who Fail to Attain the Blood Pressure Goals With Olmesartan Medoxomil 20mg Monotherapy
Brief Title: Evaluation of the Additional Efficacy, and Safety of Olmesartan Medoxomil 20mg / Hydrochlorothiazide 12.5mg in the Treatment of Chinese Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Shanghai Sankyo Pharmaceuticals Co., Ltd. (Unknown)
Responsible Party: Naotaka Ikegami, Vice President, Shanghai Sankyo Pharmaceuticals, Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SS-866 CMB/01
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Olmesartan medoxomil and hydrochlorothiazide
  Interventions: Drug: olmesartan medoxomil + hydrochlorothiazide
- 2 (Active Comparator): olmesartan medoxomil
  Interventions: Drug: olmesartan medoxomil

INTERVENTIONS:
Drug: olmesartan medoxomil + hydrochlorothiazide — olmesartan medoxomil 20mg oral tablets, once daily for 4 weeks then olmesartan medoxomil 20mg oral tablets + hydrochlorothiazide 12.5 mg oral tablets, once daily for up to 8 weeks
  Arms: 1
Drug: olmesartan medoxomil — olmesartan medoxomil 20mg oral tablets, once daily for 4 weeks then olmesartan medoxomil 40mg oral tablets, once daily for up to 8 weeks
  Arms: 2

SUMMARY:
This study is designed to evaluate the additional efficacy and safety of olmesartan medoxomil/hydrochlorothiazide in the treatment of Chinese patients with mild to moderate essential hypertension, who fail to attain the blood pressure goals with olmesartan medoxomil monotherapy

ELIGIBILITY:
Inclusion Criteria:

* At Visit 3, mean seated diastolic blood pressure (SeDBP) ≥ 95 mmHg and < 110 mmHg, AND mean seated systolic blood pressure (SeSBP) ≥140 mmHg and < 180 mmHg
* At Visit 4, mean SeDBP ≥ 90 mmH
* No significant disorder in blood, kidney, liver, cardiovascular system or endocrinology system

Exclusion Criteria:

* Patients with known or suspect secondary hypertension
* Unstable angina
* History of acute myocardial infarct, or PTCA or surgical cardiac procedures 3 months before entry into this study
* Prior or current congestive heart failure (NYHA grade III or IV), hypertrophic obstructive cardiomyopathy, valvular disease or rheumatic heart disease
* Arrhythmia of clinical significance
* Bilateral renal artery stenosis, isolated renal artery stenosis, post kidney transplantation
* Acute glomerular nephritis
* Gout sufferers, even with the normal serum uric acid at entry
* Retinal hemorrhage /exudate
* Type 1 diabetes mellitus
* Uncontrolled type 2 diabetes mellitus
* Hypovolemia
* Patients with autoimmune disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Mean change of trough seated diastolic blood pressure from baseline to Week 12 between the two treatment groups. | Baseline to12 weeks

SECONDARY OUTCOMES:
The mean change of trough seated systolic blood pressure from Week 5 to Week 12 between the two treatment groups | 8 weeks (week 5 to week 12)
The mean change of trough seated diastolic blood pressure and seated systolic blood pressure from Week 5 to Week 9 between the two treatment groups | 5 weeks (Week 5 to week 9)
The response rate in the two treatment groups from baseline to Week 9 | Baseline to 9 weeks
The response rate in the two treatment groups from baseline to Week 12 | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Naotaka Ikegami, VP, Study Director — Shanghai Sankyo Pharmaceuticals Co., Ltd.
Locations (8):
- China (8):
  - Beijing
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Wuhan